CLINICAL TRIAL: NCT03705845
Title: Actions of Dietary Tocotrienols on Obesity
Brief Title: Tocotrienols for Obesity of Postmenopausal Women
Acronym: VitE-obesity
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LBB18-147
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Postmenopausal Women
MeSH Terms: conditions — Obesity | interventions — Olive Oil; Tocotrienols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): One 430 mg olive oil softgel daily for 24 weeks. Each placebo softgel of 430 mg olive oil will contain no tocotrienol or tocopherols at detectable levels.
  Interventions: Drug: placebo softgel
- Intervention (Active Comparator): One 430 mg tocotrienol softgel daily for 24 weeks. Each tocotrienol softgel (DeltaGold® Tocotrienol 70%) contains 430 mg tocotrienol (90% δ-tocotrienol+10% γ-tocotrienol) with a 70% purity, representing 300 mg tocotrienol.
  Interventions: Drug: DeltaGold® Tocotrienol 70%

INTERVENTIONS:
Drug: placebo softgel — Each placebo softgel of 430 mg olive oil will contain no TT or tocopherols at detectable levels.
  Other Names: olive oil
  Arms: Control
Drug: DeltaGold® Tocotrienol 70% — DeltaGold® Tocotrienol 70% contains 430 mg tocotrienol (90% δ-tocotrienol + 10% γ-tocotrienol) with a 70% purity, representing 300 mg tocotrienol.
  Other Names: tocotrienols
  Arms: Intervention

SUMMARY:
Postmenopausal women are at a risk of excessive weight gain, bone loss, hypertension, and metabolic syndrome. Obesity-induced chronic low-grade inflammation is initiated by excess nutrients in metabolic cells. Recent studies have indicated tocotrienols (one kind of vitamin E, a potent antioxidant) supplement may be good for mitigating negative impacts of obesity in postmenopausal women. The purpose of the study is to examine the effect of 24-week tocotrienols on obesity-associated outcome measurements in postmenopausal women. The investigators will enroll 60 qualified women at the start of the study and randomly assigned to no tocotrienols (placebo) or tocotrienols group for 24 weeks. Obesity-associated measurements will be recorded using blood, urine, adipose tissue, and fecal samples. All data will be analyzed statistically.

DETAILED DESCRIPTION:
Postmenopausal women are at a risk of excessive weight gain, bone loss, hypertension, and metabolic syndrome. Among these risk factors, obesity is now recognized as a worldwide epidemic disease. Obesity-induced chronic low-grade inflammation is initiated by excess nutrients in metabolic cells. Aging and decline of estrogen are factors that contribute to weight gain in postmenopausal women, and approaches, such as anti-inflammatory potential in dietary antioxidants to reduce inflammation may likely combat obesity. Recent studies have indicated tocotrienols (one kind of vitamin E, a potent antioxidant) supplement may be good for mitigating negative impacts of obesity in postmenopausal women. However, no study has ever been done the role of tocotrienols in obesity-associated outcome measures in postmenopausal women. The long-term goal is to develop a new strategy featuring a dietary supplement (i.e., tocotrienols) for mitigating obesity in postmenopausal women. The purpose of the study is to examine the effect of 24-week tocotrienols on obesity-associated outcome measurements in postmenopausal women. The investigators plan to recruit postmenopausal women using flyers, non-solicited e-mail system, campus announcement, local radio, newspapers, and TV scripts. The investigators plan to enroll approximately 150-200 women to obtain 60 qualified women at the start of the study. After screening, qualified participants will be matched by body weight and age, and then randomly assigned to no tocotrienols or tocotrienols group. The outcome measures will be assessed at baseline, after 12, and after 24 weeks. Obesity-associated measurements will be recorded using blood, urine, adipose tissue, and fecal samples. The investigators will monitor safety of subjects after 12 and after 24 weeks. Food intake and physical activity will be assessed at baseline, after 12, and after 24 weeks. All data will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

1. PMW with BMI ≥30 kg/m2.
2. Normal liver, kidney, and thyroid function (TSH)-sent to Quest Diagnostic Laboratory.
3. Sedentary using International Physical Activity Questionnaire (IPAQ-short form).

Exclusion criteria

1. Unstable body weight (more than 5% change in body weight) within 3 months before intervention begins.
2. Changes to medications or supplements (i.e., steroids, statins) within 3 months of the baseline study visit that could affect lipid metabolism. • If they change any medications/supplements after the baseline visit that will affect lipid metabolism, their study participation will end.
3. Taking anticoagulants that may interact with TT.
4. Serious chronic disease (e.g., unstable cardiovascular disease, uncontrolled diabetes and hypertension, and active cancer).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Fat mass | 24 weeks
  total and regional fat mass by DXA
visceral adipose tissue | 24 weeks
  VAT by BIA

SECONDARY OUTCOMES:
total cholesterol | 24 weeks
  total cholesterol in serum
FASN | 24 weeks
  Fatty acid synthase mRNA expression in fat tissue
Oxylipins inflammation marker | 24 weeks
  oxylipins levels in plasma and adipose tissue
Gut microbiota | 24 weeks
  abundance and composition of intestinal bacteria in feces
hs-CRP | 24 weeks
  high-sensitivity C-reactive protein in serum
leptin | 24 weeks
  serum leptin
beta-oxidation | 24 weeks
  carnitine palmitoyltransferase 1A (CPT1) mRNA expression in adipose tissue
endocannabinoids inflammatory markers | 24 weeks
  endocannabinoids levels in plasma and adipose tissue
HDL | 24 weeks
  high density lipoprotein in serum
TG | 24 weeks
  triglycerides in serum

CONTACTS AND LOCATIONS:
Overall Officials: Chwan-Li Shen, PhD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aryaie A, Tinsley G, Lee J, Watkins BA, Moore L, Alhaj-Saleh A, Shankar K, Wood SR, Wang R, Shen CL. Actions of annatto-extracted tocotrienol supplementation on obese postmenopausal women: study protocol for a double-blinded, placebo-controlled, randomised trial. BMJ Open. 2020 Mar 8;10(3):e034338. doi: 10.1136/bmjopen-2019-034338. PMID 32152169